CLINICAL TRIAL: NCT05964504
Title: Improving Survival for Those With Metastatic Lobular Breast Cancer Through Development of the Multi-center PLUMB Registry-a Prospective Study of LobUlar Metastatic Breast Cancer
Brief Title: Improving Survival for Metastatic Lobular Breast Cancer (PLUMB Registry)
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 237513
Record Dates: First submitted 2023-07-19; First posted 2023-07-28 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Breast Cancer; Lobular Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Lobular | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood samples will be obtained from participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Initial Cohort: Up to 12 participants at each evaluation timepoint (approximately every 3-6 months to follow standard of care visits) will have up to 40 mL of blood drawn and distributed into 8 cell-free DNA Streck tubes, for plasma isolation, cell free DNA extraction, and ctDNA analysis. Blood for ctDNA analysis will be collected within +/- 14 days of whole body imaging studies which will occur when patients are scheduled for standard of care whole body imaging.
  Interventions: Procedure: Blood Specimen

INTERVENTIONS:
Procedure: Blood Specimen — Blood will be drawn via venipuncture

SUMMARY:
This is a prospective observational registry for patients with invasive lobular carcinoma (ILC) of the breast. After the first 1cohort is enrolled, the collected data will be utilized to develop an ILC specific response assessment tool.

DETAILED DESCRIPTION:
Primary Aims:

1. To evaluate the feasibility of developing a histologic based registry for participants living with metastatic lobular breast cancer.
2. To understand the natural history, treatment patterns, and overall survival in patients with metastatic ILC using modern, real-world data.

Secondary Aims:

1. To evaluate the correlation between imaging findings and disease progression.
2. To evaluate the correlation between ctDNA and disease progression.
3. To develop an ongoing platform for evaluating new imaging tools, tumor markers, and participant recruitment for clinical trials.

Outline:

Participants will be recruited to participate in the registry during a regularly scheduled clinic visit with their treating oncologist, and consented to participate at this time. At each evaluation time point, participants will have a blood draw performed. Participants will be followed until loss to follow up, death, or withdrawal from the registry.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed invasive lobular carcinoma. Mixed lobular/ductal cancer is allowed.
2. Age >=18 years
3. Any receptor subtype.
4. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Stage I-III breast cancer.
2. Lack of lobular histology on tumor biopsy.
3. Other active cancer (prior treated cancer with no current evidence of disease is allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with histologically proven stage IV invasive lobular carcinoma
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2034-02-28 (Estimated); Study Completion 2034-02-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility of registry | Up to 2 years
  Feasibility is defined as enrollment of 10-12 patients with metastatic ILC in the first 2 years across all participating sites, and collection of clinical assessments in >=75% of treating medical oncologists
Proportion of patients with measurable versus unmeasurable disease | Up to 10 years
  Proportion of patients with measurable disease versus unmeasurable disease using Response Evaluation Criteria in Solid Tumors (RECIST) will be reported for each line of treatment as determined by their oncologist.
Median Progression Free Survival Rate | Up to 10 years
  The median Progression-free survival rate (PFS) for participants enrolled in the registry will be utilized to develop the ILC specific response assessment tool.
Median Overall Survival Rates | Up to 10 years
  The overall rate of survival for participants enrolled in the registry will be utilized to develop the ILC specific response assessment tool.

SECONDARY OUTCOMES:
Proportion of participants who are currently taking estrogen receptor modulators or degraders | Up to 10 years
  The overall proportion of participants who are currently taking estrogen receptor modulators or degraders which may interfere with a radiolabeled form of estradiol (FES) in a positron Emission Tomography (PET) versus the participants medical oncologist assessment of disease progression will be utilized to develop the ILC specific response assessment tool.
Mean Change in Circulating tumor DNA (ctDNA) | Up to 10 years
  The overall change in quantity of ctDNA mean tumor molecules per mL blood versus medical oncologist assessment of disease progression will be utilized to develop the ILC specific response assessment tool.
Number of novel imaging tools | Up to 10 years
  The number of novel imaging tools developed during the course of data collection to improve the determination of disease status will be utilized to develop the ILC specific response assessment tool.
Number of new tumor markers introduced | Up to 10 years
  The number of participants who have detectable mutations on ctDNA evaluations with are correlated with health outcomes will be utilized to develop the ILC specific response assessment tool.
Number of participants enrolled in clinical trials | Up to 10 years
  The number of participants with metastatic ILC who have enrolled on a clinical trial will be utilized to develop the ILC specific response assessment tool.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Mukhtar, MD, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Abramson Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No